CLINICAL TRIAL: NCT05047835
Title: Comparison of Prone Position and Standard Electrocardiogram in COVID-19 Patients: A Prospective Study in Specialized COVID-19
Brief Title: Comparison of Prone Position and Standard Electrocardiogram in COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Praew Kotruchin, Associate professor, Khon Kaen University
Other Study IDs: HE641442
Record Dates: First submitted 2021-09-16; First posted 2021-09-17 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; Cardiovascular Diseases; Arrhythmias, Cardiac
Keywords: COVID-19; electrocardiogram; ARDS; Prone position
MeSH Terms: conditions — Cardiovascular Diseases; Arrhythmias, Cardiac; COVID-19 | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: electrocardiogram — Prone position electrocardiogram

SUMMARY:
Prolonged prone position ventilation reduces the 30-day mortality in acute respiratory distress syndrome (ARDS) and in COVID-19 infection.

A large number of patients with COVID-19 suffered from new-onset cardiac disease, therefore, ECG is crucial.

However, there is limited data on the effects of prone position on the ECG in COVID-19 patients.

DETAILED DESCRIPTION:
Prolonged prone position ventilation reduces the 30-day mortality in acute respiratory distress syndrome (ARDS) and in COVID-19 infection. The evidence showed that a large number of patients with COVID-19 suffered from new-onset cardiac disease due to inflammatory processes or cytokine storm, therefore, ECG is crucial for making the diagnosis including arrhythmias and myocardial infarction. However, there is limited data on the effects of prone position on the ECG in COVID-19 patients. Therefore, we aimed to identify differences of electrical parameters between prone position and standard ECG including the difference in amplitude and duration of P, QRS, PR interval, QT interval, ST-segment between both positions (supine and prone). Furthermore, we aimed to compare clinical diagnosis from EKG between prone position and standard ECG by the cardiologists.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients who were admitted to the COVID-19 specialized ward
* Age 18 -80 years old
* Suffered from pulmonary infiltration

Exclusion Criteria:

* Intubated patients
* Cardiac arrest patients whether at presentation or during the study period
* ECG cannot be performed due to anatomical defects or superficial skin problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients proved by nasal and pharyngeal swab for PCR, who were admitted to the COVID-19 specialized ward and were diagnosed with pulmonary infiltration from a chest x-ray.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of P wave amplitude | The first day of admission
  The relative changes in P-wave amplitudes with different body positions were evaluated by dividing the 12-lead ECG into subregions (I, aVL: lateral limb leads; II, III, and aVF: inferior leads; V1 to V3: anterior precordial leads; V4 to V6: lateral precordial leads).
The change of QRS-complex amplitude | The first day of admission
  The relative changes in QRS-complex amplitudes with different body positions were evaluated by dividing the 12-lead ECG into subregions (I, aVL: lateral limb leads; II, III, and aVF: inferior leads; V1 to V3: anterior precordial leads; V4 to V6: lateral precordial leads).
The change of T wave amplitude | The first day of admission
  The relative changes in T wave amplitudes with different body positions were evaluated by dividing the 12-lead ECG into subregions (I, aVL: lateral limb leads; II, III, and aVF: inferior leads; V1 to V3: anterior precordial leads; V4 to V6: lateral precordial leads).

SECONDARY OUTCOMES:
Diagnosis | The first day of admission.
  The EKG diagnosis from prone position and standard supine position which perform in the same time, in the same patient, by a cardiologist will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Khon Kaen Unversity, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: Yes
For educational or research purposes, data can be provided by contacting PI or correspondent author.
Supporting Information: Study Protocol, ICF
Time Frame: After the study finished and for 5 years later.
Access Criteria: For educational or research purposes.